CLINICAL TRIAL: NCT02165865
Title: Vascularized Composite Allotransplantation of the Hand and Upper Extremity for the Restoration of Form and Function in Hand Amputees
Brief Title: Vascularized Composite Allotransplantation of the Hand and Upper Extremity (Hand Transplant)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Illinois University (Other)
Collaborators: Memorial Medical Center Foundation (Other); Memorial Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU-SIUSOM-13-001
Record Dates: First submitted 2014-01-24; First posted 2014-06-18 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Traumatic Amputation of Arm; Traumatic Amputation of Hand
Keywords: hand transplantation; hand allotransplantation; upper extremity transplantation; upper extremity amputation; hand amputation; vascularized composite allotransplantation; composite tissue allotransplantation; variance component analysis (VCA); composite tissue allograft (CTA)
MeSH Terms: interventions — Hand Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- upper extremity/ hand transplantation (Experimental): hand transplant on unilateral dominant hand or bilateral upper extremity amputees
  Interventions: Procedure: upper extremity/ hand transplantation

INTERVENTIONS:
Procedure: upper extremity/ hand transplantation — hand transplant on unilateral dominant hand or bilateral upper extremity amputees

SUMMARY:
The Southern Illinois University (SIU) Hand Transplant Program is a multidisciplinary research effort with the goal of restoring form and function to unilateral or bilateral upper extremity amputees by vascularized composite allotransplantation of the hand/upper extremity (hand transplantation). Hand transplantation includes transferring upper extremities/hands from deceased human donors to patients with single or bilateral hand or arm amputation. The purpose of the trial is to study functional, psychological, and immunological outcomes of human upper extremity allotransplantation.

DETAILED DESCRIPTION:
Hand transplantation is the surgical attachment of a hand and sometimes an arm from an organ donor to a person who has previously suffered an amputation. It is similar to other organ transplants, such as a heart, liver, or kidney, in that the tissue comes from a deceased donor and therefore requires lifelong medications to prevent rejection. Hand transplantation also requires extensive hand rehabilitation to regain function of the transplanted limb.

The primary focus of the study is to perform hand transplantation using a steroid-sparing immunosuppression regimen, to closely follow outcomes for at least 2 years after the transplant, and to utilize new methods for immune system and functional recovery. The number and severity of side effects and the treatment provided will be analyzed in relation to the standard immunosuppressive drugs used. Functional and clinical outcomes will be correlated with data on quality of life.

After consultation with the study team and signing of the study consent forms, patients will undergo a thorough screening phase, including imaging, laboratory tests, age-appropriate screening, psychosocial evaluations, physical and occupational therapy (OT) screening, and tissue typing. Patients will then be selected by a formal patient selection committee meeting, based on results of screening procedures.

If found to be a good candidate for hand transplantation, the patient will be listed with the United Network for Organ Sharing (UNOS) to wait for a compatible donor. Organ donors from the surrounding region will be screened for compatibility in regards to blood type and tissue type, as well as hand size, skin color, tone, and hair patterns. Once a matching donor is located, the hand transplant team and participant will be notified.

After surgery the patient will stay in the intensive care unit for 1-3 days and then move to a regular hospital room where they will stay for 1-2 weeks. Physical therapy will begin within 2-3 days after surgery, and transplant staff will give daily information on the anti-rejection medications. After discharge from the hospital, the patient will stay locally for 3-6 months to monitor for signs of rejection and for extensive hand rehabilitation. Housing will be provided during this period by the hospital. Functional, psychological and immunological outcomes will then be closely followed for the life of the allograft.

ELIGIBILITY:
Inclusion Criteria:

* Recent (≥6 months) or remote (i.e., several decades) unilateral or bilateral upper limb loss from trauma or other causes desiring limb transplantation
* Below-shoulder amputation
* Male or female and of any race, color or ethnicity
* Aged 18-69 years
* Willing and able to understand and sign informed consent form
* No co-existing medical condition which, in the opinion of the study team, would place them at high risk for the surgical procedure, immunosuppression protocol, or functional results
* No co-existing psychosocial problems (i.e., alcoholism, drug abuse, lack of social support) or issue identified during psychosocial battery of testing
* Negative for malignancy for past 5 years
* Negative for hepatitis C virus or HIV at transplant
* Negative crossmatch with donor
* If female of child-bearing potential, negative serum pregnancy test
* If female of child-bearing potential, consent to use reliable contraception for at least one year following transplantation
* Willing and able to sign consents for tissue studies
* Willing to comply with Intermediate System (IS) and hand therapy protocols

Exclusion Criteria:

* Conditions that, in the opinion of the investigators, would place patient at unacceptably high risk for the surgical procedure, immunosuppression protocol, or functional results
* Sensitized recipients with high levels (>70%) of panel-reactive human leukocyte antigen (HLA) antibodies
* Conditions that may impact the success of the surgical procedure or increase the risk of postoperative complications including inherited coagulopathies like Hemophilia, Von-Willebrand's disease, Protein C and S deficiency, Thrombocythemias, Thalassemias, Sickle Cell disease, etc.
* Mixed connective tissue diseases and collagen diseases that may result in poor wound healing after surgery.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
hand allograft survival | Transplantation through end of study period (up to 5 years)

SECONDARY OUTCOMES:
hand allograft function | Transplantation through end of study period (up to 5 years)
  tests, 2 point discrimination, electromyography (EMG)/nerve conduction studies, range of motion, and a functional status assessment that includes activities of daily living
immunological response to hand transplantation | Transplantation through end of study period (up to 5 years)
  white blood cell counts, immunosuppression serum drug levels, donor specific antigen levels, tissue biopsy Banff grades
brain cortical reorganization and adaptation | Transplantation through end of study period (up to 5 years)
  functional MRI
psychosocial impact | Transplantation through end of study period (up to 5 years)
  Flannagan QOL (quality of life) survey and the Connor-Davidson Resilience Scale (CD-RISC)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Neumeister, MD, Principal Investigator — Southern Illinois University
Locations (3):
- United States (3):
  - Memorial Medical Center, Springfield, Illinois
  - SIU Institute for Plastic Surgery, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois